CLINICAL TRIAL: NCT04067518
Title: A Phase 2 Clinical Study of SHP674 in Patients With Newly Diagnosed, Untreated Acute Lymphoblastic Leukemia
Brief Title: A Clinical Study of SHP674 (Pegaspargase) in Participants With Newly Diagnosed, Untreated Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: Kyowa Kirin Co., Ltd. (Industry); ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP674-201/CL1-95014-001
Record Dates: First submitted 2019-08-13; First posted 2019-08-26 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegaspargase

STUDY DESIGN:
Intervention Model Description: The intervention study model is sequential in results section of record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SHP674 (Experimental): Part 1: Participants with ALL who were stratified into the standard risk (SR) or intermediate risk (IR) groups received total 3 doses of SHP674 in the 36-week treatment period and who were stratified into the high risk (HR) group received total 8 doses of SHP674 in the 45-week treatment period.
  Part 2: Participants with ALL who were stratified into the SR or IR groups received total 3 doses of SHP674 in the 41-week treatment period and who were stratified into the HR group received total 8 doses of SHP674 in the 45-week treatment period.
  Interventions: Biological: SHP674

INTERVENTIONS:
Biological: SHP674 — SHP674: powder for solution for injection, IV (administered by 1 to 2 hours of drip infusion), dose determination : if BSA ≥0.6 m^2: 2500 IU/m^2 every 14 days if BSA <0.6 m^2: 82.5 IU/kg every 14 days
  Other Names: Pegaspargase

SUMMARY:
The objectives of the study are to assess the safety and tolerability of a single dose of SHP674 in Japanese participants (dose confirmation) in the tolerability assessment period of Part 1 and to assess the safety, pharmacokinetics and efficacy of SHP674 dose in Part 2 (found to be tolerated in Part 1) in the treatment of newly diagnosed untreated acute lymphoblastic leukemia (ALL) in Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to ≤21 years at the time of informed consent;
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 2;
* Newly diagnosed, untreated precursor B-cell ALL
* No prior therapy for malignant tumor such as chemotherapy and radiation therapy before signing the informed consent;
* Life expectancy of at least 6 months from the date of enrollment;

Exclusion Criteria:

* Mature B-cell ALL ; Philadelphia chromosome-positive (Ph+) or BCR-ABL1-positive ALL
* Preexisting known coagulopathy ;
* History of pancreatitis;
* Continuous use of corticosteroids;
* Prior treatment or possible prior treatment with an L-asparaginase preparation;
* History of sensitivity to polyethylene glycol (PEG) or PEG-based drugs;
* Pregnant

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitose Ogawa, MD, Principal Investigator — National Cancer Center Hospital, Tokyo JAPAN
Locations (8):
- Japan (8):
  - Kagoshima University Hospital Department of Pediatrics, Kagoshima
  - Kobe Children's Hospital Department of Hematology/Oncology, Kobe
  - Nagoya Medical Center Department of Pediatrics, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Saitama Children's Medical Center Department of Hematology/Oncology, Saitama
  - Sapporo Hokuyu Hospital Department of Pediatrics and Adolescent Medicine, Sapporo
  - National Cancer Center Hospital Department of Pediatric Oncology, Tokyo
  - St. Luke's International Hospital Department of Pediatrics, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized participant-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in participants:
  * sponsored by Servier
  * with a first participant enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 8 investigative sites in Japan from 17 October 2019 to 18 January 2021. Data is reported up to primary completion date, 12 February 2021.
Pre-assignment Details: A total of 28 participants were enrolled, 3 into Part 1 and 25 into Part 2, of which 26 participants were treated, 3 in Part 1 and 23 in Part 2.
Groups:
- Part 1: SHP674: Participants with ALL who were stratified into the standard risk (SR) or intermediate risk (IR) groups received total 3 doses of SHP674, 2500 international units per square meter (IU/m^2) (if body surface area [BSA] ≥0.6 m^2) or 82.5 international units per kilogram (IU/kg) (if BSA <0.6 m^2) intravenously (IV) on Day 12 of Remission induction therapy (SR: IA2/IR: IA4) in the 5-week tolerability assessment period, Day 2 of re-induction therapy (conducted twice) in the 36-week treatment period.
- Part 2: SHP674: Participants with ALL who were stratified into the SR or IR groups received total 3 doses of SHP674, 2500 IU/m^2 (if BSA ≥0.6 m^2) or 82.5 IU/kg (if BSA <0.6 m^2) IV on Day 12 of Remission induction therapy (SR: IA2/IR: IA4), Day 2 of re-induction therapy (conducted twice) in the 41-week treatment period.
  Participants with ALL who were stratified into the HR group received total 8 doses of SHP674, 2500 IU/m^2 (if BSA ≥0.6 m^2) or 82.5 IU/kg (if BSA <0.6 m^2) IV on Day 12 of Remission induction therapy (IA4), Day 38 of early consolidation therapy, Day 6 of consolidation therapies (HR3, HR2), Day 7 of consolidation therapy (HR1), Day 2 of re-induction therapy (conducted thrice) in the 45-week treatment period.
Period: Overall Study
Arm/Group | Part 1: SHP674 | Part 2: SHP674
Started | 3 | 25
Safety Analysis Set (Safety Analysis Set (SAF) included all participants who had received at least one dose of SHP674 in Part 1 or Part 2 of the study.) | 3 | 23
- Standard Risk(SR)/Intermediate Risk (IR) | 3 | 21
- Hihg Risk (HR) | 0 | 1
- Missing | 0 | 1
Full Analysis Set (Full analysis set (FAS) included all participants who were enrolled and received SHP674 in Part 2 of the study.) | 0 | 23
Immunogenicity Analysis Set (Immunogenicity analysis set (IMAS) included all participants who had received at least one dose of SHP674 in Part 1 or Part 2 of the study and had at least one evaluable post-dose sample. If the pre-dose sample was missing it was considered negative.) | 3 | 22
Pharmacokinetic Analysis Set (Pharmacokinetic (PK) analysis included all participants enrolled in Part 1 or Part 2 who had received first dose of SHP674 at remission induction therapy, who were evaluable for non-compartmental analysis and included only the participants who had sufficient samples collected to provide interpretable PK results with no deviations that might had affected the PK interpretation.) | 3 | 23
Completed | 2 | 20
Not Completed | 1 | 5
Not completed — Adverse Event | 1 | 3
Not completed — Screen failures | 0 | 1
Not completed — Enrolled but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: SAF included all participants who had received at least one dose of SHP674 in Part 1 or Part 2 of the study.
Groups:
- Part 1: SHP674: Participants with ALL who were stratified into the SR or IR groups received total 3 doses of SHP674, 2500 IU/m^2 (if BSA ≥0.6 m^2) or 82.5 IU/kg (if BSA <0.6 m^2) IV on Day 12 of Remission induction therapy (SR: IA2/IR: IA4) in the 5-week tolerability assessment period, Day 2 of re-induction therapy (conducted twice) in the 36-week treatment period.
- Part 2: SHP674: Participants with ALL who were stratified into the SR or IR groups received total 3 doses of SHP674, 2500 IU/m^2 (if BSA ≥0.6 m^2) or 82.5 IU/kg (if BSA <0.6 m^2) IV on Day 12 of Remission induction therapy (SR: IA2/IR: IA4), Day 2 of re-induction therapy (conducted twice) in the 41-week treatment period and who were stratified into the HR group received total 8 doses of SHP674, 2500 IU/m^2 (if BSA ≥0.6 m^2) or 82.5 IU/kg (if BSA <0.6 m^2) IV on Day 12 of Remission induction therapy (IA4), Day 38 of early consolidation therapy, Day 6 of consolidation therapies (HR3, HR2), Day 7 of consolidation therapy (HR1), Day 2 of re-induction therapy (conducted thrice) in the 45-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Part 1: SHP674 | Part 2: SHP674 | Total
Number analyzed (Participants) | 3 | 23 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.63) | 6.7 (4.79) | 7.1 (4.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 1 | 12 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Definition of racial groups according to NIH (National Institutes of Health) and OMB (Office of Management and Budget)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 3 | 23 | 26
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 23 | 26

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and SHP-674-Related TEAEs During the Tolerability Assessment Period
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant after signing informed consent. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease, whether or not it is related to the investigational product. TEAE is defined as any untoward medical occurrence in a participant who received an investigational product which occurs during the period from Day 1 of the pre-treatment phase to 30 (+7) days after the last dose of investigational product, or until the start of a new therapy, whichever occurs first. A related adverse event signifies that there is a reasonable causal relationship between study treatment and an AE.
Time Frame: Up to 30 days after last dose of study drug (approximately 49 weeks)
Population: SAF (Safety Analysis Set) included all participants who had received at least one dose of SHP674 in Part 1 or Part 2 of the study. As pre-specified in the protocol, this outcome measure is analyzed only for Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: SHP674
Number analyzed (Participants) | 3
Participants
  TEAEs | 3
  SHP-674-Related TEAEs | 3

2. Primary Outcome: Part 2: Percentage of Participants Who Achieved a Plasma Asparaginase Activity of ≥0.1 International Units Per Milliliter (IU/mL) 14 Days (336 Hours) After the First Dose of SHP674
Time Frame: 14 days after the first dose of SHP674
Population: FAS (Full Analysis Set) included all participants who were enrolled and received SHP674 in Part 2 of the study.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Part 2: SHP674
Number analyzed (Participants) | 23
participants | 100.0 [85.2 to 100.0]

3. Secondary Outcome: Percentage of Participants With Anti-Drug (SHP674) Antibody (ADA) (Part 1 and Part 2)
Time Frame: Predose and 25 days post dose (Part 1 and Part 2)
Population: Immunogenicity analysis set (IMAS) included all participants who had received at least one dose of SHP674 in Part 1 or Part 2 of the study and had at least one evaluable post-dose sample. If the pre-dose sample was missing it was considered negative.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: SHP674 | Part 2: SHP674
Number analyzed (Participants) | 3 | 22
Participants
  Pre-existing ADA positive | 0 | 4
  Seroconversion upon tretament | 0 | 2

4. Secondary Outcome: Percentage of Participants With Anti-Polyethylene Glycol (PEG) Antibody (Part 1 and Part 2)
Time Frame: Predose and 25 days post dose (Part 1 and part 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: SHP674 | Part 2: SHP674
Number analyzed (Participants) | 3 | 22
Participants
  Pre-existing Anti-PEG positive | 0 | 2
  Seroconversion upon treatment | 0 | 0

5. Secondary Outcome: Part 1: Percentage of Participants Who Achieved a Plasma Asparaginase Activity of ≥0.1 IU/mL 14 Days (336 Hours) After the First Dose of SHP674
Time Frame: 14 days after the first dose of SHP674
Population: SAF included all participants who had received at least one dose of SHP674 in Part 1 or Part 2 of the study. As pre-specified in the protocol, this outcome measure is analyzed only for Part 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1: SHP674: Participants with Acute Lymphoblastic Leukemia (ALL) who were stratified into the SR or IR groups received total 3 doses of SHP674, 2500 IU/m^2 (if BSA ≥0.6 m^2) or 82.5 IU/kg (if BSA <0.6 m^2) IV on Day 12 of Remission induction therapy (SR: IA2/IR: IA4) in the 5-week tolerability assessment period, Day 2 of re-induction therapy (conducted twice) in the 36-week treatment period.
Arm/Group | Part 1: SHP674
Number analyzed (Participants) | 3
percentage of participants | 100.0 [29.2 to 100.0]

6. Secondary Outcome: Part 2: Percentage of Participants With Plasma Asparaginase Activity of ≥0.1 IU/mL or <0.1 IU/mL
Time Frame: Day 1 (pre-dose, 5 min, 4 hours, 24 hours post dose), Days 2, 4, 11, 14, 18, 25 post dose
Population: FAS included all participants who were enrolled and received SHP674 in Part 2 of the study. Number analyzed indicates the number of participants analyzed at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: SHP674
Number analyzed (Participants) | 23
percentage of participants
  ≥0.1 IU/mL: Day 1 (pre-dose) | 0.0 [0.0 to 14.8]
  ≥0.1 IU/mL: Day 1 (5 mins post dose): number analyzed (Participants) | 22
  ≥0.1 IU/mL: Day 1 (5 mins post dose) | 100.0 [84.6 to 100.0]
  ≥0.1 IU/mL: Day 1 (4 hours post dose) | 100.0 [85.2 to 100.0]
  ≥0.1 IU/mL: Day 1 (24 hours post dose) | 100.0 [85.2 to 100.0]
  ≥0.1 IU/mL: Day 2 post dose | 100.0 [85.2 to 100.0]
  ≥0.1 IU/mL: Day 4 post dose | 100.0 [85.2 to 100.0]
  ≥0.1 IU/mL: Day 11 post dose | 100.0 [85.2 to 100.0]
  ≥0.1 IU/mL: Day 14 post dose | 100.0 [85.2 to 100.0]
  ≥0.1 IU/mL: Day 18 post dose: number analyzed (Participants) | 22
  ≥0.1 IU/mL: Day 18 post dose | 95.5 [77.2 to 99.9]
  ≥0.1 IU/mL: Day 25 post dose: number analyzed (Participants) | 22
  ≥0.1 IU/mL: Day 25 post dose | 50.0 [28.2 to 71.8]
  <0.1 IU/mL : Day 1 (pre-dose) | 100.0 [85.2 to 100.0]
  <0.1 IU/mL: Day 1 (5 mins post dose): number analyzed (Participants) | 22
  <0.1 IU/mL: Day 1 (5 mins post dose) | 0.0 [0.0 to 15.4]
  <0.1 IU/mL: Day 1 (4 hours post dose) | 0.0 [0.0 to 14.8]
  <0.1 IU/mL: Day 1 (24 hours post dose) | 0.0 [0.0 to 14.8]
  <0.1 IU/mL: Day 2 post dose | 0.0 [0.0 to 14.8]
  <0.1 IU/mL: Day 4 post dose | 0.0 [0.0 to 14.8]
  <0.1 IU/mL: Day 11 post dose | 0.0 [0.0 to 14.8]
  <0.1 IU/mL: Day 14 post dose | 0.0 [0.0 to 14.8]
  <0.1 IU/mL: Day 18 post dose: number analyzed (Participants) | 22
  <0.1 IU/mL: Day 18 post dose | 4.5 [0.1 to 22.8]
  <0.1 IU/mL: Day 25 post dose: number analyzed (Participants) | 22
  <0.1 IU/mL: Day 25 post dose | 50.0 [28.2 to 71.8]

7. Secondary Outcome: Survival Rate at 1 Year After the Start of Study Treatment
Description: Survival rate is defined as the percentage of subjects who survived at 1 year after the start of study treatment.
Time Frame: 1 year after the start of study treatment (from first dose up to 12 months)
Population: The analysis was performed on the safety set analysis, defined as the set of all subjects who had received at least one dose of SHP674 in Part 1 or Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: SHP674 | Part 2: SHP674
Number analyzed (Participants) | 3 | 23
Participants | 3 | 23

8. Secondary Outcome: Event-free Survival Rate at 1 Year After the Start of Study Treatment
Description: Event-free survival rate is defined as percentage of subjects who did not experience any event and survived at 1 year after the start of study treatment.
Time Frame: 1 year after the start of study treatment (from first dose up to 12 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: SHP674 | Part 2: SHP674
Number analyzed (Participants) | 3 | 23
Participants | 3 | 23

ADVERSE EVENTS:
Time Frame: Parts 1 and 2: Up to 30 days after last dose of study drug (approximatively 117 weeks)
Description: SAF included all participants who had received at least one dose of SHP674 in Part 1 or Part 2 of the study. As planned and pre-specified in protocol, the safety data was analyzed for Part 1 and Part 2 of study.
Arm/Group | Part 1: SHP674 | Part 2: SHP674
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/3 | 10/23
Other Adverse Events (participants affected / at risk) | 3/3 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: SHP674 (N=3) | Part 2: SHP674 (N=23)
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: SHP674 (N=3) | Part 2: SHP674 (N=23)
Anaemia (Blood and lymphatic system disorders) | 3 | 21
Coagulopathy (Blood and lymphatic system disorders) | 0 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 18
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 | 4
Cushingoid (Endocrine disorders) | 1 | 5
Blepharitis (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 2
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Anal erosion (Gastrointestinal disorders) | 0 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 17
Dental caries (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 10
Gastric haemorrage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Hypoasthesia oral (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 14
Proctalgia (Gastrointestinal disorders) | 1 | 2
Proctitis (Gastrointestinal disorders) | 0 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 13
Vomiting (Gastrointestinal disorders) | 2 | 18
Catheter site erythema (General disorders) | 2 | 1
Catheter site pain (General disorders) | 1 | 3
Chilis (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 0
Hunger (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 11
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 9
Hepatic steatosis (Hepatobiliary disorders) | 1 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 7
Seasonal allergy (Immune system disorders) | 0 | 2
Bacteriaemia (Infections and infestations) | 1 | 4
Conjunctivitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 10
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 4
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 2
Procedural headache (Injury, poisoning and procedural complications) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 5
Alanine aminotransferase increased (Investigations) | 0 | 13
Amylase increased (Investigations) | 0 | 3
Antithrombin III decreased (Investigations) | 3 | 12
Antithrombin III increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 13
Blood albumin decreased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 3 | 9
Blood cholesterol increased (Investigations) | 1 | 3
Blood fibrinogen decreased (Investigations) | 3 | 16
Blood fibrinogen increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 2
Blood urea increased (Investigations) | 1 | 2
C-reactive protein increased (Investigations) | 0 | 2
Coagulation test abnormal (Investigations) | 0 | 2
Fibrin D dimer increased (Investigations) | 2 | 1
Fibrin degradation products increased (Investigations) | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 9
Immunoglobulins decreased (Investigations) | 0 | 4
Liver function test abnormal (Investigations) | 2 | 1
Liver function test increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 6
Neutrophil count decreased (Investigations) | 0 | 7
Plasmin inhibitor decreased (Investigations) | 3 | 3
Plasminogen decreased (Investigations) | 3 | 3
Platelet count decreased (Investigations) | 3 | 21
Protein total decreased (Investigations) | 2 | 1
Weight decreased (Investigations) | 0 | 2
Weight increased (Investigations) | 0 | 4
White blood cell count decreased (Investigations) | 3 | 21
Central obesity (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 8
Increased appetite (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholinergic syndrome (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 11
Leukoencephalopathy (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Taste disorder (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 1 | 1
Depressive symptom (Psychiatric disorders) | 0 | 3
Discouragement (Psychiatric disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 6
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 3
Calculus urinary (Renal and urinary disorders) | 1 | 1
Glycosuria (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive sough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 17
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 10
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04067518/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT04067518/SAP_001.pdf